CLINICAL TRIAL: NCT02116465
Title: Open-label, Two-treatment, 4-period Replicated Crossover Study in Healthy Subjects to Investigate the Plasma Pharmacokinetics of Levodopa and Carbidopa After Oral Administration of Single Doses of Two Fixed-dose Combination Products
Brief Title: Pharmacokinetic Study With Levodopa-carbidopa Fixed-dose Products in Healthy Subjects After Oral Administration
Acronym: LCD18K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LCD-018/K; 2013-003175-35 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Fasted State
MeSH Terms: conditions — Fasting | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Levodopa Carbidopa 100/25 tablets Test 1 (Active Comparator): single oral dose of levodopa carbidopa immediate release tablets
  Interventions: Drug: Levodopa Carbidopa immediate release tablets
- Levodopa Carbidopa 100/25 tablets Ref. 1 (Active Comparator): single oral dose of levodopa carbidopa immediate release tablets
  Interventions: Drug: Levodopa Carbidopa immediate release tablets
- Levodopa Carbidopa 100/25 tablets Test 2 (Active Comparator): single oral dose of levodopa carbidopa immediate release tablets
  Interventions: Drug: Levodopa Carbidopa immediate release tablets
- Levodopa Carbidopa 100/25 tablets Ref. 2 (Active Comparator): single oral dose of levodopa carbidopa immediate release tablets
  Interventions: Drug: Levodopa Carbidopa immediate release tablets

INTERVENTIONS:
Drug: Levodopa Carbidopa immediate release tablets — oral administration
  Other Names: isicom 100/25 mg; Nacom 100/25 mg

SUMMARY:
The study is carried-out to describe and compare the plasma pharmacokinetics of levodopa and carbidopa after oral single-dose administration of 100 mg levodopa plus 25 mg carbidopa by means two fixed combination products (test: Isicom® 100/25 mg; reference: Nacom® 100/25 mg).

Additionally, to describe and compare the safety and tolerability of the two investigational treatments administered to healthy subjects.

DETAILED DESCRIPTION:
Isicom® 100/25 mg and Sinemet® (Trade name in Germany: Nacom®) 100/25 mg are authorised fixed-combination products containing 100 mg levodopa plus 25 mg carbidopa. These two formulations were tested for bioequivalence in 1997 (DESITIN trial № LCD-010/K); based on the regulatory provisions in place at that time (CPMP/EWP/QWP/1401/98), the two formulations could be accepted to be bioequivalent.

The present study is proposed to be conducted in order to verify and confirm the bioequivalence of Isicom® 100/25 mg (test formulation) and Nacom® 100/25 mg (reference formulation) in agreement with the pertinent regulatory guidance that came in place 2010 (CHMP Guideline On The Investigation Of Bioequivalence - CPMP/EWP/QWP/1401/98- Rev. 1/ Corr - Jan.2010).

ELIGIBILITY:
Inclusion Criteria:

* Males or females (females of non-childbearing potential or of childbearing potential while taking medically appropriate contraception)
* Race: Caucasian
* Age: 18 to 45 years
* Body weight: 50 100 kg
* Body Mass Index: 18 26 kg.m-2
* Healthy based on the screening examination
* Willing and able to provide informed consent

Exclusion Criteria:

* Previous participation in this trial or participant in any other trial during the last 90 days
* Donation of blood or plasma during the last 90 days or a history of blood loss exceeding 300 mL within the last 3 months
* History of any clinically relevant allergy including hypersensitivity to levodopa or carbi-dopa and related excipients
* Presence of any acute or chronic infection
* Presence or history of any relevant co-morbidity
* Resting systolic blood pressure > 160 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
* Clinically relevant ECG-abnormalities, in particular prolonged QTc(F) of > 450 msec in males and > 460 msec in females
* Presence of any relevant abnormality in the laboratory safety tests, especially low haemo-globin (< 120 g/L in females and (< 136 g/L in males) and increased liver enzymes (2 times the upper limit of the normal range)
* Positive serology for HBsAg or anti HCV
* Positive HIV test
* Positive alcohol or urine drug test at screening
* Regular use of any prescription medicine (except for contraceptives) or over-the-counter product, herbal product, hormone supplement, etc. in the 30 days prior to the Screening visit
* History of alcohol and/or drug abuse and/or daily use of > 30 g alcohol
* Smoking more than 10 cigarettes/day or equivalent of other tobacco products
* Suspicion or evidence that the subject is not trustworthy and reliable
* Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard.
* Positive pregnancy test
* Lactating
* Female subjects of child-bearing potential not using appropriate contraception in the 3 weeks prior to enrolment until two weeks after the last dose of the trial medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cmax and AUC(0-tz) of levodopa and carbidopa | 12 hours
  Cmax (maximal plasma concentration), AUC (area under the curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Sofia, Bulgaria